CLINICAL TRIAL: NCT06656130
Title: Comparative Effects of Pranayama and Jacobson;s Progressive Muscle Relaxation Technique on Cardiovascular Parameters,Stress and Quality of Life in Pre-hypertension
Brief Title: Pranayama and Jacobson's Progressive Muscle Relaxation Technique in Pre-hypertensive Patients
Acronym: PRANvsJPMR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huma52160
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Prehypertension
Keywords: : Jacobson's Progressive Muscle Relaxation Technique, Pranayama, Pre-hypertension
MeSH Terms: conditions — Prehypertension | interventions — Respiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of Pranayama on cardiovascular parameters, stress and quality of life in pre-hypertension (Experimental): This group will receive Pranayama. Pranayama is the practice of breath regulation. It's a main component of yoga, an exercise for physical and mental wellness. The practice of pranayama involves breathing exercises and patterns. You purposely inhale, exhale, and hold your breath in a specific sequence. Interventions will be performed for 30 minutes in a day, 3 days per week for 8 weeks. (total no. of sessions=24). Breathing exercises will be consist on Alternate Nostril Technique, Skull Shinning Technique, Bellow Breath, Bee Breath, Victorious Breath
  Interventions: Other: Pranayama
- effects of Jacobson's technique on CVS parameters, stress and QOL in Pre-hypertension (Experimental): This group will receive Jacobson's Progressive Muscle Relaxation Technique. Jacobson's relaxation technique is a type of therapy that focuses on tightening and relaxing specific 14 muscle groups in sequence. It's also known as progressive relaxation therapy. By concentrating on specific areas and tensing and then relaxing them, you can become more aware of your body and physical sensations, The sessions will consist of 30 minutes in a day, 3 days per week for 8 weeks. (total no. of sessions=24).
  Interventions: Other: Jacobson's progressive muscle relaxation technique

INTERVENTIONS:
Other: Pranayama — Pranayama is the practice of breath regulation. It's a main component of yoga, an exercise for physical and mental wellness. The practice of pranayama involves breathing exercises and patterns. Patient purposely inhale, exhale, and hold his/her breath in a specific sequence.
  Other Names: Breathing Technique
  Arms: Effects of Pranayama on cardiovascular parameters, stress and quality of life in pre-hypertension
Other: Jacobson's progressive muscle relaxation technique — Jacobson's relaxation technique is a type of therapy that focuses on tightening and relaxing specific 14 muscle groups in sequence. It's also known as progressive relaxation therapy. By concentrating on specific areas and tensing and then relaxing them, patient can become more aware of his/her body and physical sensations,
  Other Names: Breathing and stretching technique
  Arms: effects of Jacobson's technique on CVS parameters, stress and QOL in Pre-hypertension

SUMMARY:
Objective of our study is to determine the comparative effects of Pranayama and Jacobson's Relaxation Technique on cardiovascular parameters, stress and quality of life in Pre-hypertensive patients.

This study is used to determine the effects of Pranayama versus Jacobson's Progressive Muscle Relaxation Technique on cardiorespiratory parameters, stress and quality of life in pre-hypertensive patients.

This randomized clinical trial (RCT) endeavors to enroll ___ participants, divided equally into Pranayama and Jacobson's Progressive Muscle Relaxation Technique groups. The non-probability convenient sampling technique, followed by random allocation using a lottery method, ensures a diverse yet unbiased sample. Study is being conducted at the Kashmir Medical Complex Sialkot.

The Pranayama group(n=25) undergoes sessions three times a week, emphasizing breathing techniques like alternate nostril technique and bellow breathing.

The Jacobson's Progressive Muscle Relaxation Technique group(n=25) follows a similar schedule, engaging in full-body relaxation exercises targeting major muscle groups. Parameters will be assessed on 1st day, 3rd week and 8th week by outcome measures, SPSS version 23 will be used for analysis.

DETAILED DESCRIPTION:
This is a randomized controlled trial used to determine the effects of Pranayama and Jacobson's progressive muscle relaxation technique on Cardiovascular parameters, Stress and Quality of Life in Prehypertensive Patients.

A Nonprobability Convenient Sampling Technique will be used and random allocation into groups using the Lottery method. Patients will be assigned into 2 groups i.e. Group A & Group B Group A: will receive Pranayama. Pranayama is the practice of breath regulation. It's a main component of yoga, an exercise for physical and mental wellness. The practice of pranayama involves breathing exercises and patterns. Patient will purposely inhale, exhale, and hold his/her breath in a specific sequence. Interventions will be performed for 30 minutes in a day, 3 days per week for 8 weeks. (total no. of sessions=24). Breathing exercises will be consist on Alternate Nostril Technique, Skull Shinning Technique, Bellow Breath, Bee Breath, Victorious Breath Group B: will receive Jacobson's Progressive Muscle Relaxation Technique. Jacobson's relaxation technique is a type of therapy that will focus on tightening and relaxing specific 14 muscle groups in sequence. It's also known as progressive relaxation therapy. By concentrating on specific areas and tensing and then relaxing them, Patient can become more aware of his/her body and physical sensations, The sessions will consist of 30 minutes in a day, 3 days per week for 8 weeks. (total no. of sessions=24).

Prior to the study, all participants will be informed of the purpose and method of conducting the research. Each of them will sign an informed consent to participate in the study and to process personal data for scientific purposes. We confirm that all research will be performed in accordance with relevant guidelines and regulations.

Participants will be divided into 2 experimental groups. Group 1 will perform Pranayama and Group 2 will perform Jacobson's progressive muscle relaxation technique.

Both the interventions will be performed for 30 minutes in a day, 3 days per week for 8 weeks.

SPSS for Windows software, version 25 will be used to analyze the data using statistical significance p=0.05. After assessing the normality, if the p-value is greater than 0.05, a parametric test will be applied. If the p-value is less than 0.05 then a nonparametric test will be applied.

Descriptive Statistics: Frequency tables, pie charts, and bar charts will be used for categorical data to show a summary of group measurements measured over time.

Difference between groups: Anova Test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 30 and 60 years old.
* Gender: Male and Female both.
* Diagnosed patients of Pre-hypertension.
* Stable health condition to participate in moderate physical activities.
* Willing to comply with the study protocol, including attending scheduled exercise sessions and follow-up assessments

Exclusion Criteria:

* Diagnosed case of Hypertension or takes any antihypertensive medication.
* Patient having any other associated systemic disorder are excluded.
* Severe physical limitations, disabilities, or musculoskeletal disorders.
* History of substance abuse.
* Patients with Neurological diseases
* Patients with severe or unstable heart conditions, recent heart attack, or heart failure, other cardiovascular disorders

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
PSR (Perceived Stress Scale) | 8 weeks
  The Perceived Stress Scale (PSS) is one of the most widely used instruments to measure stress perceptions. The original PSS is a 14-item self-report measure designed to assess "the degree to which situations in one's life are appraised as stressful". It is a global measure of stress, rather than a measure of specific stressful life events. Specifically, items assess the extent to which one's life is perceived as "unpredictable, uncontrollable, and overloading
SF-12 (QOL) | 8 weeks
  Quality of life (QOL) is a broad multidimensional concept that usually includes subjective evaluations of both positive and negative aspects of life. The SF-12 Health Survey version 2 (SF-12v2) is a generic short-form health survey developed in the USA from the original SF36. It produces two summary measures evaluating physical and mental self-perceived health; for this reason, it could be a suitable and complete tool to assess the self-perceived quality of life of university students because it allows investigating both the aspects

CONTACTS AND LOCATIONS:
Overall Officials: Sumera AbdulHameed Supervisor/ Research Incharge, M.PHIL, Principal Investigator — Riphah International University Lahore
Locations (1):
- Sialkot Medical and Physiotherapy Center, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No